CLINICAL TRIAL: NCT02760823
Title: Alpha Lipoic Acid as an Adjuvant Treatment in Acute Phosphide Poisoning: A Randomized Clinical Trial
Brief Title: Alpha Lipoic Acid as an Adjuvant Treatment in Acute Phosphide Poisoning
Acronym: ALA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heba Allah Ali Abd El-Halim Mabrouk (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Heba Allah Ali Abd El-Halim Mabrouk, Principal Investigator, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALA-2016-CT; ALA (Registry Identifier: Alpha Lipoic Acid)
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Toxicity
MeSH Terms: interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha Lipoic Acid (Active Comparator): Subjects in this arm will receive ALA IV, as a dose of 600 mg/12 hours.
  Interventions: Drug: Alpha Lipoic Acid (Thioctacid)
- Non-Alpha Lipoic Acid (Placebo Comparator): Subjects in this arm will to receive standard treatment only (without Alpha Lipoic Acid, instead they will receive placebo , which is determined by the attending physician who maintains clinical responsibility for all patients. It consists of patient resuscitation, gastric decontamination (with sodium bicarbonate, and activated charcoal [1 g/Kg, orally] in the first 6 hours after onset of poisoning), adequate hydration and supportive treatment.
  Interventions: Drug: Placebo (for Alpha Lipoic Acid)

INTERVENTIONS:
Drug: Alpha Lipoic Acid (Thioctacid) — 600 mg/12 hours, IV (in the vein)
  Other Names: Thioctic Acid
  Arms: Alpha Lipoic Acid
Drug: Placebo (for Alpha Lipoic Acid) — Normal saline in syringe simulating Alpha Lipoic Acid 600mg
  Arms: Non-Alpha Lipoic Acid

SUMMARY:
The aim of this study is to evaluate efficacy and safety of Alpha Lipoic Acid(ALA) as an adjuvant in the management of patients with acute phosphide poisoning.

DETAILED DESCRIPTION:
The study will be carried out following approval of the research ethical committee of Tanta Faculty of Medicine on patients admitted to The Poison Control Unit (Emergency Hospital, Tanta University and Emergency Hospital, Mansoura University) with acute phosphide poisoning in the period from January 2016 to January 2018. A written informed consent will be taken from each patient or his/her guardians (if the patient was unable to participate in the consent process). Confidentiality of the data will be maintained by making code numbers for each patient. The investigators plan to conduct a randomized clinical trial to evaluate efficacy and safety of ALA as an adjuvant in treatment of patients with acute phosphide poisoning. Fifty patients will be randomized to ALA or a non ALA in a 1:1 ratio (25 patients in each group). ALA will be given IV, as a dose of 600 mg/12 hours. Patients will be monitored and a detailed documentation of any adverse effect due to ALA therapy will be recorded.

This intervention represents an added treatment to the existing standard of care. All patients will continue to receive standard treatment, which is determined by the attending physician who maintains clinical responsibility for all patients. It consists of patient resuscitation, gastric decontamination (with sodium bicarbonate, and activated charcoal [1 g/Kg, orally] in the first 6 hours after onset of poisoning), adequate hydration and supportive treatment. All the patients will be followed up until discharge or death. All patients will be subjected to:

I. History. II. Clinical examination. III. Laboratory investigations: At admission and repeated before discharge.

ELIGIBILITY:
Inclusion Criteria:

Patients (male or female, aged 12 years or older) with symptomatic acute phosphide poisoning (deliberate or accidental), with diagnosis made on the basis of:

1. The typical clinical manifestations due to and following shortly after a single exposure to phosphide.
2. Reliable identification of the compound based on the container brought by patient attendants or a subsequent confirmation by silver nitrate test for phosphine detection in stomach contents.

Exclusion Criteria:

* Patients less than 12 years of age
* Pregnant and lactating women
* Patients with ingestion or exposure to other substances in addition to phosphide.
* Patients with other major medical conditions (e.g. cardiovascular disease, renal or hepatic failure).
* Patients presenting more than 6 hours of having consumed the phosphide compound (late presenters).
* Patients treated for acute phosphide poisoning in any medical center before admission.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  Death Rate

SECONDARY OUTCOMES:
Duration of hospital stay | 2 years
  Duration that patient will stay in hospital

OTHER OUTCOMES:
Need for intubation | 2 years
  will the patient need to be intubated or not